CLINICAL TRIAL: NCT03657368
Title: Ventilation Strategy During General Anesthesia for Orthopedic Surgery: A Quality Improvement Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 18-001
Record Dates: First submitted 2018-08-31; First posted 2018-09-05 (Actual); Results first posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-02

CONDITIONS: Orthopedic Surgery; Ventilation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low tidal volume and low PEEP (Experimental): Ventilation parameters will be set at tidal volume = 6 ml/ kg predicted body weight, and PEEP = 5 cm water (H2O).
  Interventions: Procedure: Low tidal Volume; Procedure: Low PEEP
- Low tidal volume and high PEEP (Experimental): Ventilation parameters will be set at tidal volume = 6 ml/kg predicted body weight, and PEEP = 8 cm H2O.
  Interventions: Procedure: Low tidal Volume; Procedure: High PEEP
- High tidal volume and low PEEP (Experimental): Ventilation parameters will be set at tidal volume = 10 ml/kg predicted body weight, and PEEP = 5cm H2O.
  Interventions: Procedure: High tidal Volume; Procedure: Low PEEP
- High tidal volume and high PEEP (Experimental): Ventilation parameters will be set at tidal volume = 10 ml/kg predicted body weight, and PEEP = 8cm H2O.
  Interventions: Procedure: High tidal Volume; Procedure: High PEEP

INTERVENTIONS:
Procedure: Low tidal Volume — Tidal volume = 6 ml/kg predicted body weight
  Arms: Low tidal volume and high PEEP; Low tidal volume and low PEEP
Procedure: High tidal Volume — Tidal volume = 10 ml/kg predicted body weight
  Arms: High tidal volume and high PEEP; High tidal volume and low PEEP
Procedure: Low PEEP — PEEP = 5 cm H2O
  Arms: High tidal volume and low PEEP; Low tidal volume and low PEEP
Procedure: High PEEP — PEEP = 8 cm H2O
  Arms: High tidal volume and high PEEP; Low tidal volume and high PEEP

SUMMARY:
The objective is to determine the optimal intraoperative ventilation strategy among the chosen tidal volume and positive end-expiratory pressure (PEEP) levels, and standardize it in an enhanced recovery pathway for orthopedic surgical patients. In particular, we propose to determine which combination of intraoperative tidal volume and positive end-expiratory pressure is best for patients having elective orthopedic surgery.

DETAILED DESCRIPTION:
This is a non-randomized alternating intervention cohort study in which all orthopedic surgery operating rooms will alternate amongst four designated ventilation settings which include two tidal volumes and two PEEP levels. At the end of the four-week sequence, the entire sequence will be repeated 26 times over a 2-year period. Thus, ventilator settings will not be randomized on a per-patient basis, or even among study weeks.

Ventilation parameters will be designated at the beginning of each study week. However, clinicians will be free to adjust to whatever ventilation settings they believe is optimal in individual patients to ensure oxygenation and patient safety.

ELIGIBILITY:
Inclusion Criteria:

* Surgery in orthopedic operating rooms 32-37
* General anesthesia with endotracheal intubation.

Exclusion Criteria:

* Non-orthopedic procedures;
* Intubation before induction of anesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2860 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alparslan Turan, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared on a collaborative basis.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication of the primary manuscript.
Access Criteria: Data will be shared on a collaborative basis with investigators who plan substantive sub-analyses.

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Tidal Volume and Low PEEP: Ventilation parameters will be set at tidal volume = 6 ml/ kg predicted body weight, and PEEP = 5 cm water (H2O). (n = 727)
  Low tidal Volume: Tidal volume = 6 ml/kg predicted body weight
  Low PEEP: PEEP = 5 cm H2O
- Low Tidal Volume and High PEEP: Ventilation parameters will be set at tidal volume = 6 ml/kg predicted body weight, and PEEP = 8 cm H2O. (n = 635)
  Low tidal Volume: Tidal volume = 6 ml/kg predicted body weight
  High PEEP: PEEP = 8 cm H2O
- High Tidal Volume and Low PEEP: Ventilation parameters will be set at tidal volume = 10 ml/kg predicted body weight, and PEEP = 5cm H2O. (n = 799)
  High tidal Volume: Tidal volume = 10 ml/kg predicted body weight
  Low PEEP: PEEP = 5 cm H2O
- High Tidal Volume and High PEEP: Ventilation parameters will be set at tidal volume = 10 ml/kg predicted body weight, and PEEP = 8cm H2O. (n = 699)
  High tidal Volume: Tidal volume = 10 ml/kg predicted body weight
  High PEEP: PEEP = 8 cm H2O
Period: Overall Study
Arm/Group | Low Tidal Volume and Low PEEP | Low Tidal Volume and High PEEP | High Tidal Volume and Low PEEP | High Tidal Volume and High PEEP
Started | 727 | 635 | 799 | 699
Completed | 727 | 635 | 799 | 699
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Tidal Volume and Low PEEP | Low Tidal Volume and High PEEP | High Tidal Volume and Low PEEP | High Tidal Volume and High PEEP | Total
Number analyzed (Participants) | 727 | 635 | 799 | 699 | 2860
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (15) | 64 (14) | 62 (15) | 63 (14) | 63 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 360 | 326 | 442 | 376 | 1504
  Male | 367 | 309 | 357 | 323 | 1356
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  race: White | 603 | 511 | 655 | 575 | 2344
  race: Black | 97 | 108 | 115 | 89 | 409
  race: other | 16 | 12 | 15 | 22 | 65
  race: missing | 11 | 4 | 14 | 13 | 42
BMI [Mean (Standard Deviation); unit: kg/m2] | 30 (7) | 30 (7) | 31 (8) | 32 (7) | 31 (7)
ASA score [Count of Participants; unit: Participants] — The ASA score refers to the American Society of Anesthesiologists (ASA) Physical Status Classification System, which is used to assess the preoperative physical health of a patient before surgery. ASA score and measure description:
  I: A normal, healthy patient. II: A patient with mild systemic disease. III: A patient with severe systemic disease. IV: A patient with severe systemic disease that is a constant threat to life. V: A moribund patient who is not expected to survive without the operation. VI: A declared brain-dead patient whose organs are being removed for donor purposes.
  Participants
    1 | 23 | 9 | 10 | 14 | 56
    2 | 122 | 106 | 157 | 120 | 505
    3 | 519 | 460 | 572 | 520 | 2071
    4 or 5 | 63 | 60 | 60 | 45 | 228
The total Charlson score [Median (Inter-Quartile Range); unit: units on a scale] — The Charlson Comorbidity Index (CCI), it is a weighted score used to predict the risk of mortality or adverse outcomes by assessing the presence of various comorbid conditions (chronic diseases or medical conditions).
  Each condition is assigned a specific weight (from 1 to 6 points) based on the associated risk of mortality. e.g. Dementia scored 1, Metastatic solid tumor scored 6. The total Charlson score is the sum of the CCI for all conditions that a patient has. A higher score indicates a higher risk of death or complications due to the comorbidities. The range is 0 to 37 or higher.
  units on a scale | 1 [0 to 2] | 1 [0 to 2] | 1 [0 to 2] | 1 [0 to 2] | 1 [0 to 2]
smoking [Count of Participants; unit: Participants] | 369 | 346 | 404 | 341 | 1460
COPD [Count of Participants; unit: Participants] | 87 | 85 | 103 | 102 | 377
Obstructive sleep apnea [Count of Participants; unit: Participants] | 161 | 144 | 202 | 187 | 694
Asthma [Count of Participants; unit: Participants] | 119 | 105 | 157 | 102 | 483
intraoperative use of Rocuronium [Median (Inter-Quartile Range); unit: mg] | 70 [50 to 90] | 70 [50 to 90] | 70 [50 to 90] | 65 [50 to 90] | 68 [50 to 90]
Crystalloids [Mean (Standard Deviation); unit: L] | 1.7 (0.8) | 1.7 (0.8) | 1.8 (0.8) | 1.7 (0.8) | 1.7 (0.8)
blood loss [Median (Inter-Quartile Range); unit: ml] | 150 [50 to 300] | 150 [50 to 250] | 200 [50 to 300] | 150 [50 to 300] | 150 [50 to 300]
transfusion [Count of Participants; unit: Participants] | 48 | 50 | 75 | 50 | 223

OUTCOME MEASURES:

1. Primary Outcome: Time-weighted Average SaO2/FiO2 Ratio in the Postanesthesia Care Unit (PACU)
Description: Primary outcome was oxygenation in the postoperative care unit, defined by the peripheral oxygen saturation divided by the fraction of inspired oxygen (SpO2/FiO2 ratio), a validated measure of acute lung injury.
Time Frame: After surgery until discharged from PACU or up to 90 minutes
Population: The mean difference was estimated from a linear mixed regression model with surgeries from same patient as repeated measures, after propensity score weighting.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- TV = 6 ml/kg: tidal volume = 6 ml/kg
- TV = 10 ml/kg: tidal volume = 10 ml/kg
- PEEP = 5cmH2O: Positive End-Expiratory Pressure = 5cmH2O
- PEEP = 8cmH2O: Positive End-Expiratory Pressure = 8cmH2O
Arm/Group | TV = 6 ml/kg | TV = 10 ml/kg | PEEP = 5cmH2O | PEEP = 8cmH2O
Number analyzed (Participants) | 1362 | 1498 | 1526 | 1334
ratio | 355 (46) | 350 (47) | 353 (46) | 352 (47)
Statistical Analysis 1: Comparison: TV = 6 ml/kg vs TV = 10 ml/kg; Test type: Superiority; p = 0.042, Regression, Linear; Mean Difference (Final Values) = 3.5, 97.5% CI 2-sided [-0.4 to 7.3]
Statistical Analysis 2: Comparison: PEEP = 5cmH2O vs PEEP = 8cmH2O; Test type: Superiority; p = 0.966, Regression, Linear; Mean Difference (Final Values) = -0.1, 97.5% CI 2-sided [-3.9 to 3.7]

2. Secondary Outcome: Composite of Serious Postoperative Pulmonary Complications
Description: Postoperative diagnoses will be collected from electronic medical records of patients. Individual chart reviews (blinded to ventilation management) will confirm that terms of the composite are met will be performed.
Time Frame: After surgery from 2 to 5 days
Measure: Number; unit: person
Groups:
- PEEP = 5cmH2O: PEEP = 5cmH2O
- PEEP = 8cmH2O: PEEP = 8cmH2O
Arm/Group | TV = 6 ml/kg | TV = 10 ml/kg | PEEP = 5cmH2O | PEEP = 8cmH2O
Number analyzed (Participants) | 1362 | 1498 | 1526 | 1334
person | 34 | 39 | 36 | 37
Statistical Analysis 1: Comparison: TV = 6 ml/kg vs TV = 10 ml/kg; Test type: Superiority; p = 0.519, Regression, Logistic; Odds Ratio (OR) = 0.93, 99.2% CI 2-sided [0.68 to 1.27]
Statistical Analysis 2: Comparison: PEEP = 5cmH2O vs PEEP = 8cmH2O; Test type: Superiority; p = 0.232, Regression, Logistic; Odds Ratio (OR) = 0.87, 99.2% CI 2-sided [0.63 to 1.19]

3. Secondary Outcome: Oxygenation in Ward, Defined as Time Weighted Average (TWA) of SaO2/FIO2 Ratio
Description: Oxygen administration and SaO2 are normally recorded at 4-hour intervals on surgical wards. The time weighted average (TWA) of overall SaO2/FIO2 ratio will be compared among different ventilation strategies.
Time Frame: After surgery from 2 to 5 days
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | TV = 6 ml/kg | TV = 10 ml/kg | PEEP = 5cmH2O | PEEP = 8cmH2O
Number analyzed (Participants) | 1362 | 1498 | 1526 | 1334
ratio | 428 (42) | 430 (41) | 429 (41) | 429 (41)
Statistical Analysis 1: Comparison: TV = 6 ml/kg vs TV = 10 ml/kg; Test type: Superiority; p = 0.217, Regression, Linear; Mean Difference (Final Values) = -2.1, 99.2% CI 2-sided [-6.5 to 2.4]
Statistical Analysis 2: Comparison: PEEP = 5cmH2O vs PEEP = 8cmH2O; Test type: Superiority; p = 0.660, Regression, Linear; Mean Difference (Final Values) = 0.7, 99.2% CI 2-sided [-3.7 to 5.2]

4. Secondary Outcome: Length of Postoperative Hospital Stay by Days
Description: The days of postoperative hospitalization, which from out of operation room to discharge from the hospital, an average of 1 week
Time Frame: from out of operation room to discharge
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | TV = 6 ml/kg | TV = 10 ml/kg | PEEP = 5cmH2O | PEEP = 8cmH2O
Number analyzed (Participants) | 1362 | 1498 | 1526 | 1334
days | 3 [2 to 5] | 3 [2 to 5] | 3 [2 to 5] | 3 [2 to 5]
Statistical Analysis 1: Comparison: TV = 6 ml/kg vs TV = 10 ml/kg; Test type: Superiority; p = 0.143, Mixed Models Analysis; mean ratio = 1.03, 99.2% CI 2-sided [0.97 to 1.10]
Statistical Analysis 2: Comparison: PEEP = 5cmH2O vs PEEP = 8cmH2O; Test type: Superiority; p = 0.649, Regression, Logistic; mean ratio = 0.99, 99.2% CI 2-sided [0.93 to 1.05]

5. Other Pre Specified Outcome: Patients Need of Oxygen in Ward After Surgery
Description: number of patients who need of Oxygen in ward after surgery during hospital stay
Time Frame: from out of operation room to discharge from the hospital
Measure: Number; unit: participants
Groups:
- PEEP = 5cmH2O: Positive End-Expiratory Pressure= 5cmH2O
Arm/Group | TV = 6 ml/kg | TV = 10 ml/kg | PEEP = 5cmH2O | PEEP = 8cmH2O
Number analyzed (Participants) | 1362 | 1498 | 1526 | 1334
participants | 855 | 932 | 961 | 826

6. Other Pre Specified Outcome: Patients With Unplanned ICU Admission
Description: number of patients with unplanned ICU admission after surgery in hospital stay
Time Frame: from out of operation room to discharge from the hospital
Measure: Number; unit: participants
Arm/Group | TV = 6 ml/kg | TV = 10 ml/kg | PEEP = 5cmH2O | PEEP = 8cmH2O
Number analyzed (Participants) | 1362 | 1498 | 1526 | 1334
participants | 44 | 43 | 43 | 44

ADVERSE EVENTS:
Time Frame: 1 week.
Description: None observed
Groups:
- Low Tidal Volume and Low PEEP: tidal volume = 6 ml/kg and PEEP = 5 cmH2O
- High Tidal Volume and Low PEEP: tidal volume = 10 ml/kg and PEEP = 5 cmH2O
- Low Tidal Volume and High PEEP: tidal volume = 6 ml/kg and PEEP = 8 cmH2O
- High Tidal Volume and High PEEP: tidal volume = 10 ml/kg and PEEP = 8 cmH2O
Arm/Group | Low Tidal Volume and Low PEEP | High Tidal Volume and Low PEEP | Low Tidal Volume and High PEEP | High Tidal Volume and High PEEP
All-Cause Mortality (participants affected / at risk) | 0/727 | 0/635 | 0/799 | 0/699
Serious Adverse Events (participants affected / at risk) | 0/727 | 0/635 | 0/799 | 0/699
Other Adverse Events (participants affected / at risk) | 0/727 | 0/635 | 0/799 | 0/699

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/68/NCT03657368/Prot_SAP_000.pdf